CLINICAL TRIAL: NCT04394494
Title: A Randomized Clinical Trial of Extension for Low Back Pain: Motor Imagery of Extension Versus Physical Extension Exercises
Brief Title: RCT of Motor Imagery of Extension for LBP vs. Exercise
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: St. Ambrose University (Other)
Responsible Party: Principal Investigator, Kevin Farrell, Professor and Chair, Orthopaedic Residency Program in Physical Therapy, St. Ambrose University
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Treatment
Other Study IDs: SAU McKenzie MI
Record Dates: First submitted 2020-05-14; First posted 2020-05-19 (Actual); Last update posted 2022-05-26 (Actual); Status verified 2022-05

CONDITIONS: Low Back Pain
Keywords: Motor Imagery; McKenzie; Low Back Pain; Directional preference
MeSH Terms: conditions — Low Back Pain

STUDY DESIGN:
Intervention Model Description: This is an Randomized Control Trial. Subjects with LBP will be allocated to one of 2 study groups.
Who Masked: Participant
Masking Description: Patients will be assigned in an alternating order to either the experimental or control group.
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Motor Imagery (Experimental): Patients are instructed in a motor imagery protocol of imaging extension exercises (similar to the CG), without doing the actual extension exercises. Patients will be instructed in visualizing them moving into extension and back as well as common sensations they may experience (as if doing the actual exercise). They will repeat the visualization process 10 times while in the clinic, after which they will be instructed in a home program containing the same treatment - every 2 hours, perform 10 visualization exercises.
  Interventions: Other: Motor Imagery. Imaging doing Extension exercises without actually doing them.
- Control (Active Comparator): Patients are instructed in extension exercises and actually, physically doing the actual extension exercises. Patients will physically repeat the extension exercises 10 times while in the clinic, after which they will be instructed in a home program containing the same treatment - every 2 hours, perform 10 exercises.
  Interventions: Other: Control: Physically performing extension based exercises.

INTERVENTIONS:
Other: Motor Imagery. Imaging doing Extension exercises without actually doing them. — This study will compare imagining doing specific extension based exercises for LBP vs. actually performing the exercises. This intervention will be just imaging doing the exercises.
  Arms: Motor Imagery
Other: Control: Physically performing extension based exercises. — This study will compare imagining doing specific extension based exercises for LBP vs. actually doing them. This intervention will be actually, physically performing the exercises.
  Arms: Control

SUMMARY:
Low back pain (LBP) is the most common musculoskeletal condition treated in physical therapy, accounting for an estimated 25-40% of outpatient physical therapy visits. One strategy commonly used for treating LBP is directional preference. Directional preference is the process of examining a patient with LBP's response to a movement direction, i.e., extension, and if it coincides with improvement, the test becomes part of the treatment. Various studies have shown evidence for, and use of directional preference by physical therapists. Specifically for LBP, directional preference usually involves either an extension-bias or flexion-bias, with various studies indication an extension protocol being the most common (estimated > 80% of patients). With extension exercises, a favorable therapeutic effect result in centralization of symptoms (leg pain migrates proximal), improved range of motion (ROM), decreased pain and decreased fear of movement.

In recent years there has been an increased interest in various pain neuroscience strategies to help people in pain, including LBP. It is well established that the physical body of a person is represented in the brain by a network of neurons, often referred to as a representation of that particular body part in the brain. This representation refers to the pattern of activity that is evoked when a particular body part is stimulated. The most famous area of the brain associated with representation is the primary somatosensory cortex (S1). These neuronal representations of body parts are dynamically maintained. It has been shown that patients with pain display different S1 representations than people with no pain. The interesting phenomenon associated with cortical restructuring is the fact that the body maps expand or contract, in essence increasing or decreasing the body map representation in the brain. Furthermore, these changes in shape and size of body maps seem to correlate to increased pain and disability. Various studies have shown that physical movement is associated with restoring the cortical maps, which in turn may be associated with a decreased pain experience.

In patients with high levels of pain, sensitization of the nervous system and fear of movement, physical movement itself may increase a pain experience. An added therapeutic ability to help restore these cortical maps is motor imagery (visualization). Various studies have shown that motor imagery activate the same areas of the brain as when actually physically moving, thus restoring the altered maps "without moving."

DETAILED DESCRIPTION:
* Patient arrive to physical therapy with low back pain (physician referral or self-referral)
* Patient complete standard clinic medical and insurance intake forms
* Based on the intake forms, patients are screened by the physical therapists against the inclusion criteria and if met, asked to participate in the study
* Upon agreement, a written consent is signed
* Patients complete research intake forms:

  * Demographic information
* Age
* Gender
* Duration of LBP
* Location of LBP (body chart with grid allocation)

  * Pain rating (NPRS): Numeric Pain Rating Scale
  * Fear-Avoidance (Physical and Work Subscales) (FABQ)
  * Pain Catastrophization Scale (PCS)
* Patients undergo a standard physical therapy interview
* Patients undergo a standard physical therapy examination
* Patients undergo a directional preference test to determine if they are potentially responsive to extension exercises
* Once patients are shown to be responsive to extension, they are alternately allocated to receive motor imagery of extension exercises (experimental group; [EG]) or physical extension exercises (control group, [CG]).
* Prior to the treatment lumbar extension ROM will be measured via a standardized procedure
* Upon completion of the tests, patients will receive one of two allocated treatments

Following the treatment, patients will undergo repeat measures of:

* Spinal extension ROM
* Pain rating
* Fear of movement
* Pain catastrophization Patients will be asked to return to physical therapy in 2 to 3 days (standard care)

Upon return, measurements will be repeated of:

* Pain rating
* Fear of movement
* Pain catastrophization
* Spinal extension ROM This marks the end of data collection (and study) of the individual patient - Following the tests the patient is treated per the discretion of the therapist as the data collection has been completed

ELIGIBILITY:
Inclusion Criteria:

* LBP of less than 3 months duration
* Age 18-65
* Able to read and understand English
* Fit directional preference of extension

Exclusion Criteria:

* Any red flags for therapy
* Prior spinal surgery
* Directional preference of flexsion

Ages: 18 Years to 65 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 10 (Actual)
Dates: Start 2019-05-25 (Actual); Primary Completion 2020-08-01 (Actual); Study Completion 2020-08-30 (Actual)

PRIMARY OUTCOMES:
Spine ROM | within a single, 90 minute session
  range patient is able to bend backward
Pain rating | within a single, 90 minute session
  Numeric pain rating Scale 0 - 10 (0 = no pain and 10 = worst pain). The minimal detectable change (MDC) for the NPRS for low back pain is reported to be 2.0.
Fear of Movement | within a single, 90 minute session
  Fear Avoidance Belief Questionnaire (FABQ): The FABQ is a self-report of patients feelings about their fear to move.
Pain Catastrophization | within a single, 90 minute session
  Pain Catastrophization Scale: The PCS is a self-report questionnaire assessing inappropriate coping strategies and catastrophic thinking about pain and injury. on a 13-item, 5-point Likert scale with higher scores indicating elevated levels of catastrophizing.

CONTACTS AND LOCATIONS:
Overall Officials: Kevin Farrell, Principal Investigator — St. Ambrose University
Locations (4):
- United States (4):
  - Edward Elmhurst Health Physical Therapy, Naperville, Illinois
  - Kevin Farrell, Davenport, Iowa
  - Rock Valley Physical Therapy, Davenport, Iowa
  - Genesis Physical Therapy - 53rd St, Davenport, Iowa

IPD SHARING:
Plan to Share IPD: No
There are no plans to share any of individual's data. All data will be coded for data entry and analysis by research team.